CLINICAL TRIAL: NCT02358746
Title: Ventricular Tachycardia in Ischemic Cardiomyopathy; a Combined Endo-Epicardial Ablation Within the First Procedure Versus a Stepwise Approach a Randomized Controlled Trial
Brief Title: Ventricular Tachycardia in Ischemic Cardiomyopathy; a Combined Endo-Epicardial Ablation Within the First Procedure Versus a Stepwise Approach
Acronym: EPILOGUE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Astrid Hendriks, MD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL48168.078.14
Record Dates: First submitted 2015-01-27; First posted 2015-02-09 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Ventricular Tachycardia; Ischemic Cardiomyopathy
Keywords: epicardial catheter ablation
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combined endo/epicardial approach (Experimental): combining endocardial scar homogenization with epicardial scar homogenization in the first VT ablation approach
  Interventions: Other: combined endo/epicardial approach
- stepwise approach (Active Comparator): endocardial scar homogenization only at the first VT ablation procedure
  Interventions: Other: stepwise approach

INTERVENTIONS:
Other: combined endo/epicardial approach
  Other Names: endo /epicardial catheter ablation
  Arms: combined endo/epicardial approach
Other: stepwise approach — endocardial scar homogenization only at the first VT ablation procedure
  Arms: stepwise approach

SUMMARY:
Rationale: Nowadays ventricular tachycardia (VT) ablation in structural heart disease is performed primarily by early referral; while at the same time we still struggle with the limited longterm ablation success of endocardial VT ablation. An underestimated number of VTs from ischemic substrate have an epicardial exit. However, one cannot accurately predict who is in need of epicardial ablation. The investigators hypothesise endo/epicardial substrate homogenization in a first approach to be superior to endocardial substrate homogenization alone, in terms of recurrence on follow-up.

Objective: To show superiority of a combined endo/epicardial approach compared to a stepwise approach in the ablation of ventricular tachycardia in a population with ischemic cardiomyopathy on VT recurrence.

Study design: Multicenter prospective open randomized controlled trial. Study population: All patients above 18 years with an ischemic cardiomyopathy being referred for a ventricular tachycardia ablation.

Intervention: One group undergoes endo/epicardial ablation and the other group has endocardial ablation only as a first approach.

Main study parameters/endpoints: The main study endpoint is the difference in recurrences of ventricular tachycardia on follow-up - clinical or on implantable cardioverter defibrillator (ICD) interrogation - between the two ablation groups; secondary endpoints are procedure success and safety.

ELIGIBILITY:
Inclusion Criteria:

1. clinical indication for ablation of a monomorphic ventricular tachycardia referred to one of the participating ablation centers
2. history of ischemic heart disease
3. ICD carrier or ICD implantation planned after the ablation
4. informed written consent

Exclusion Criteria:

1. current unstable angina as defined by current european guidelines
2. AMI < 30 days or in case of incessant VT < 14 days
3. absence of visualisation of the coronary anatomy (coronary angiogram /CT-angiogram)
4. significant coronary stenosis approachable and clinically relevant for intervention
5. presence of a mobile left ventricle thrombus seen on (contrast) echocardiography or MRI
6. previous pericarditis
7. presence of mitral/aortic mechanical valves prosthesis; previous coronary artery bypass graft; any other thoracic surgery that could cause pericardial adhesions
8. previous thoracic radiation therapy
9. contra-indication for general anaesthesia
10. age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2015-05; Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence (Recurrence of any ventricular tachycardia) | 2 years
  Recurrence of any ventricular tachycardia: any appropriate ICD therapy or VT > 30 seconds of duration recorded by ICD interrogations or on clinical event recorded by electrocardiogram with an initial blanking period of 1 week after the ablation procedure

SECONDARY OUTCOMES:
procedure success | 2 years
  success: non-inducibility of any sustained monomorphic VT partial success: non-inducibility of clinical VT (inducibility of non-clinical VT excluding polymorphic VT, VT with cycle length < 200ms)
procedure related (serious) adverse events | 30 days
  major: death, acute myocardial infarction (AMI) / coronary artery damage, major bleeding - type III and V, abdominal bleeding, tamponade > 80cm3, late tamponade, ischemic cerebral event minor: dry right ventricle puncture, drainable hemopericardium, postprocedural precordial pain, phrenic nerve injury, minor bleeding - type II
procedure time, fluoroscopy and radiofrequency time | one day
time to recurrence to ventricular arrhythmia | 2 years
number of appropriate ICD therapy on follow-up | 2 years
number of ventricular arrhythmia related hospitalizations | 2 years
free of antiarrhythmic drugs on follow-up | 2 years
repeat procedure | 2 years
incessant VT or VT storm on follow-up | 2 years
mortality | 2 years